CLINICAL TRIAL: NCT06282536
Title: Neoadjuvant Therapy With Iruplinalkib for Potentially Resectable ALK Positive Non-Small Cell Lung Cancer: A Single Arm, Exploratory Trial
Brief Title: Neoadjuvant Therapy With Iruplinalkib for Potentially Resectable ALK Positive NSCLC: A Single Arm, Exploratory Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Director, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-018
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Potentially Resectable ALK Positive Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; ALK; Iruplinalkib; Potentially Resectable Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: All enrolled patients received Iruplinalkib neoadjuvant therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Therapy With Iruplinalkib (Experimental): In this arm, 20 patients with III-IVA stage, potentially resectable ALK Positive non-small cell lung cancer will receive 4 circles of neoadjuvant Iruplinalkib. And the patients who are resectable after neoadjuvant therapy will be treated with surgery. Postoperative patients receive adjuvant Iruplinalkib therapy up to 2 years/until the disease progressed.
  Interventions: Drug: Iruplinalkib; Procedure: surgery

INTERVENTIONS:
Drug: Iruplinalkib — 60 mg on days 1-7, if tolerable, 180 mg from day 8 onwards.
Procedure: surgery — Patients with resectable tumors after neoadjuvant therapy will be treated with surgery.

SUMMARY:
Fusion of anaplastic lymphoma kinase (ALK) is an important driving gene for NSCLC, with an incidence rate of 3-7%. In patients with advanced ALK mutation NSCLC, first-line use of ALK inhibitors significantly improves progression free survival. The perioperative research on ALK positive NSCLC was relatively late, and currently most studies mainly focus on early to mid stage ALK positive NSCLC patients. The results of two Phase III clinical trials showed that second-generation ALK targeted drugs, neoadjuvant and/or adjuvant therapy for ALK positive NSCLC, significantly prolonged DFS in patients, including increased pathological response rate, median response duration, and prolonged OS. For ALK positive advanced NSCLC patients who are resistant to second-generation ALK targeted drugs, there is currently limited exploration and there is an urgent need for new exploratory clinical studies.This trial aims to evaluate the effectiveness of Iruplinalkib neoadjuvant therapy for potentially resectable ALK positive non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient shall sign the Informed Consent Form. 2.Aged 18 ≥ years. 3.Histological or cytological diagnosis of NSCLC by needle biopsy, and evaluated by researchers as stage III-IVA, and diagnosed as ALK positive through genetic testing.

  4.Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1. 5. According to the MDT evaluation (which should include a thoracic surgeon specializing in tumor surgery), it is considered that the primary NSCLC is potentially completely resectable; 6. At least 1 measurable lesion according to RECIST 1.1. 7.Patients with good function of other main organs (liver, kidney, blood system, etc.) 8.Patients with lung function can tolerate surgery; 9.Fertile female patients must voluntarily use effective contraceptives not less than 120 days after chemotherapy or the last dose of toripalimab (whichever is later) during the study period, and urine or serum pregnancy test results within 7 days prior to enrollment are negative. 10. Unsterilized male patients must voluntarily use effective contraception during the study period not less than 120 d

Exclusion Criteria:

* 1. Previously received targeted therapy (including TKI or monoclonal antibodies), immunotherapy, or any investigational drug treatment for NSCLC; 2.Pathological confirmation of mixed small cell and non-small cell lung cancer; 3.Patients with a malignancy other than NSCLC within five years prior to the start of this trial，except for cured basal cell carcinoma of the skin, early gastrointestinal (GI) carcinoma excised through endoscopy, cervical carcinoma in situ, ductal carcinoma in situ of the breast, papillary thyroid carcinoma, or any cured cancer deemed to have no impact on the survival of the current NSCLC; 4.Participants with any unstable systemic disease (including active infection, uncontrolled hypertension), unstable angina pectoris, angina pectoris starting in the last three months, congestive heart failure (>= NYHA) Grade II), myocardial infarction (6 months before admission), severe arrhythmia requiring drug treatment, liver, kidney or metabolic diseases; 5.Patients with congenital or acquired immune dysfunction (such as HIV infected individuals); 6.Received other major surgical treatments (excluding diagnosis) within 4 weeks prior to the start of the study or expected to undergo major surgical treatments during the study period; 7.Participants who are allergic to the test drug or any auxiliary materials; 8.A history of extensive diffuse bilateral interstitial fibrosis in the past or before medication, or a known grade 3 or 4 history of interstitial fibrosis or interstitial lung disease, including pneumonia, allergic pneumonia, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, and pulmonary fibrosis, but not including local radiation pneumonia or radiation pulmonary fibrosis history;8. Pregnant or lactating women; 9.Any malabsorption; 10.Participants suffering from nervous system diseases or mental diseases that cannot cooperate 11.Other factors that researchers think it is not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 30 months
  ORR is defined according to the RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Pathologic complete response (PCR) rate | Up to 30 months
  PCR rate is defined as the proportion of participants who have achieved pathologic complete response (on routine hematoxylin and eosin staining, no tumor cell can be found in tumor bed or lymph node) in all participants.
Major pathologic response (MPR) rate | Up to 30 months
  MPR rate is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants.
Overall survival (OS) | up to 60 months
  It is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
Event-free survival (EFS) | up to 60 months
  Event-free survival (EFS) is defined as the length of time (months) from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Treatment-related adverse event (TRAE) | Up to 30 months
  TRAE is defined and classified according to NCI-CTCAE v5.0 in all participants.
5-year overall survival (OS) | Up to 72 months
  OS is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
1-year event-free survival (EFS) rate | Up to 24 months
  Event-free survival (EFS) is defined as the length of time (months) from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note:
  the appearance of one or more new lesions is also considered progression).
Health related quality of life (HRQol) | Up to 36 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30 & LC13, Version 3). EORTC's QLQ-C30 & LC13 (V3.0) is a core scale for lung cancer patients, with a total of 43 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options. The other items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published.